CLINICAL TRIAL: NCT00470782
Title: Changes in Aerobic Capacity and Body Composition in Colon Cancer Patients Receiving Chemotherapy
Brief Title: Aerobic Capacity and Body Composition in Colon Cancer Patients
Status: Completed | Type: Observational
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: GI-5-0064 / ethics 23429
Record Dates: First submitted 2007-05-07; First posted 2007-05-08 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2012-04

CONDITIONS: Colonic Neoplasms
Keywords: colonic neoplasms; exercise; body composition; anthropometry
MeSH Terms: conditions — Colonic Neoplasms; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Recent studies have shown that survival after a colorectal cancer diagnosis may be affected by a person's activity level and body size. This research says that for colorectal cancer patients, the less active and more obese they are, the more likely they are to have a cancer recurrence or die from their cancer. Chemotherapy has been shown to reduce activity levels, fitness, and body size in some cancer patients. However, it is not known how chemotherapy specific for colon cancer patients affects their activity levels, fitness, and body size. The main goal of our study will be to look at how chemotherapy treatments affect the fitness, activity levels, and body size in colon cancer patients. In order to do this, we will measure these variables before chemotherapy treatments, and at 1 and 6 months following the end of treatment. Our results will show how chemotherapy affects fitness, activity levels, and body size in colon cancer patients and provide data to help in designing an exercise intervention specifically for colon cancer survivors.

DETAILED DESCRIPTION:
Background Information: Recent evidence has suggested that the physical activity levels and body composition of colorectal cancer survivors can impact the disease-free and overall survival following diagnosis, with those individuals who are more overweight or obese and less active at greater risk of a recurrence of or dying from colorectal cancer (Meyerhardt et al, 2006a,b; Digman et al, 2006). Chemotherapy treatments have been shown to improve survival in a number of cancer populations, but unfortunately they have also been shown to negatively impact numerous physiological and psychological variables, including reduced exercise capacity, self-reported physical functioning and activity levels, and negative changes in body composition (Schmitz et al, 2005). This suggests that chemotherapy treatments may negatively impact variables that have been associated with survival in individuals diagnosed with colorectal cancer. However, this research has been conducted in cancer populations other than colorectal cancer patients, hence the specific impact of the chemotherapy treatments for colorectal cancer on these outcomes is not known.

Objectives: The primary objective of the study is to determine the effects of chemotherapy treatments on the aerobic capacity and body composition of colon cancer patients. Secondary objectives are to determine the effects of chemotherapy treatments on quality of life, fatigue, performance status, self-reported and objectively measured physical functioning, exercise behaviour, oxygen uptake kinetics, muscular strength, and anthropometric variables.

Study Design: The study parameters assessed will include descriptive information on demographic, lifestyle and medical variables; a graded exercise test with metabolic measurement to determine peak oxygen consumption (VO2peak); air-displacement plethysmography (BOD POD) testing and anthropometric measurements (waist & hip circumferences, waist-to-hip ratio, body mass index) to assess body composition; a questionnaire to determine cancer-specific quality of life and fatigue (Functional Assessment of Cancer Treatment - Colorectal and Fatigue); performance status assessment (Eastern Cooperative Oncology Group performance status); self-reported (Medical Outcomes Study Short Form-36 Physical Function Scale) and objectively measured (Physical Functional Performance-10 and Senior's Fitness Tests) physical functioning; self-reported exercise behavior (Godin Leisure Time Exercise Questionnaire); submaximal exercise test with metabolic measurement to determine oxygen uptake kinetics; an 8-repetition maximum test to assess upper (bench press) and lower (leg press) body muscular strength; and a fasted blood sample to be used for future biomarkers assays. All of these assessments will be completed at baseline prior to the subject's first chemotherapy infusion, and 1 and 6 months after the completion of all chemotherapy infusions.

The following calculation was used to estimate the required sample size based on the primary outcome of aerobic capacity (Peak Oxygen Consumption; VO2peak): n = 2 + C (s/d)2 (Snedecor et al, 1989), where C is a constant equal to 7.85 for a power of 0.80 and alpha of 0.05, s is the standard deviation of 6.0 ml/kg/min, and d is a 3.5 ml/kg/min difference between groups. Therefore, a sample size of 25 subjects is required to detect a 1 Metabolic Equivalent (MET) or 3.5 ml/kg/min reduction in VO2peak in colorectal cancer survivors following the completion of chemotherapy treatment, with a standard deviation (SD) in oxygen consumption of 6.0 ml/kg/min, a power of 0.80, and an alpha set at p<0.05 (two-tailed). Each 1 MET change in exercise capacity has been positively associated with a 12% difference in overall survival in the general population (Myers et al, 2002). A sample of 30 subjects will be recruited to account for any subjects lost to follow-up. To compare the effects of chemotherapy treatment on the study assessments to colon cancer surgery alone, 10 subjects will be recruited to complete all of the study assessments at the same 3 time points to allow for a "surgery only" comparison group.

Inclusion/Exclusion Criteria: Inclusion criteria will include: 1)histologically confirmed colon cancer (Stage III and those Stage II patients deemed high-risk 2) approval of the treating oncologist 3) they will receive chemotherapy 4) able to understand and provide written informed consent in English 5) 18+ years of age 6) no uncontrolled co-morbidities (including hypertension, cardiac illness, psychiatric condition, etc.) negative ECG as assessed during maximal graded exercise test *Ten patients meeting all eligibility requirements except for criteria 3 will be recruited to the study to serve as "surgery only" controls.

Exclusion criteria include 1) metastatic or recurrent colon cancer patients; 2) pregnancy; 3) any uncontrolled medical condition that would be a contraindication to exercise (assessed by treating oncologist); 4) unwilling to attend, travel to, or participate in the assessments at all 3 time points.

Recruitment: Patients will be recruited from outpatient colorectal clinics at the Cross Cancer Institute. The project coordinator will be present at all clinics, and in conjunction with the treating oncologist and clinic nurses will screen patient lists to determine eligibility for that day. The treating medical oncologist will have final determination of patient eligibility for the study and will introduce the trial to the patient if they are deemed to meet all eligibility requirements. If the patient expresses interest, he or she will be approached by the project coordinator who will discuss the study in further detail and will also give the patient a study information package. The patient will be told that a follow-up phone call will be made in the next few days to confirm if the patient is interested in participating in the trial. If the patient is still interested, all baseline testing appointments will be scheduled. Based on an estimate of 8 new colon cancer patients eligible for the study in clinic per week and a 15% accrual rate, it should take approximately 36 weeks to recruit the required number of subjects (n = 30).

Statistical Analysis: Data will be analyzed using SPSS version 15.0 software (SPSS, Inc., Evanston, IL). The principal analyses of end points will employ the last observation carried forward approach. Independent t-tests will be used to test for variables differentiating between patients accepting/declining participation and completing/dropping out of study. Descriptive statistics will be used to summarize all study assessment data at each time point. The changes in measured outcomes from baseline to post-chemotherapy (4 weeks post) to recovery (24 weeks post-chemotherapy) will be analysed using a one-way analysis of variance for repeated measures. Any differences in study outcomes between subjects receiving chemotherapy versus those who are receiving surgery alone will be analysed using a two-way analysis of variance for repeated measures.

Stopping Rules: Subjects are free to withdraw from the study at any time, which includes stopping at any point during any of the study assessments.

Data Safety Monitoring Committee: Ethical and scientific approval will be obtained from Alberta Cancer Board and the Health Ethics Research Board at the University of Alberta. All data will be number coded so that the identity of participants cannot be traced. All data will be kept in a secure, locked cabinet in the Behavioral Medicine Laboratory and will only be accessible to members of the research team. The local Institutional Research Ethics Boards will oversee the validity and integrity of data by conducting periodic audits of study records.

The safety of participants will be of primary concern at all times. Study investigators will monitor participants during all study assessments. All adverse events, however minor, will be recorded. All serious adverse events will be reported to the local Institutional Research Ethics Boards, as well as each participant's treating oncologist. The project coordinator, under the supervision of the principal investigator, will be responsible for reporting any serious adverse events.

References:

Dignam JJ, Polite BN, Yothers G, Raich P, Colangelo L, O'Connell MJ, Wolmark N. (2006). Body mass index and outcomes in patients who receive adjuvant chemotherapy for colon cancer. Journal of the National Cancer Institute. 98:1647-1654.

Meyerhardt JA, Giovannucci EL, Holmes MD, Chan AT, Chan JA, Colditz GA, Fuchs CS. (2006a). Physical activity and survival after colorectal cancer diagnosis. Journal of Clinical Oncology. 24:3527-3534.

Meyerhardt JA, Heseltine D, Niedzwiecki D, Hollis D, Saltz LB, Mayer RJ, Thomas J, Nelson H, Whitton R, Hantel A, Schilsky RL, Fuchs CS. (2006b). Impact of physical activity on cancer recurrence and survival in patients with stage III colon cancer: findings from CALGB 89803. Journal of Clinical Oncology. 24:3535-3541.

Schmitz KH, Holtzman J, Courneya KS, Masse LC, Duval S, Kane R. (2005). Controlled physical activity trials in cancer survivors: a systematic review and meta-analysis. Cancer Epidemiology, Biomarkers & Prevention. 14:1588-1595.

Snedecor G, Cochran W, Cox D. (1989). Statistical Methods (8th ed). The Iowa State University Press.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed colon cancer (Stage III and those Stage II patients deemed high-risk
* approval of the treating oncologist
* scheduled to received chemotherapy
* able to understand and provide written informed consent in English
* 18+ years of age
* no uncontrolled co-morbidities (including hypertension, cardiac illness, psychiatric condition, etc.)
* negative ECG as assessed during maximal graded exercise test

Exclusion Criteria:

* metastatic or recurrent colon cancer patients
* pregnancy
* any uncontrolled medical condition that would be a contraindication to exercise (assessed by treating oncologist)
* unwilling to attend, travel to or participate in the assessments at all 3 time points

In addition, 10 patients meeting all of the eligibility criteria who are not scheduled to receive chemotherapy will also be recruited to the study to serve as "surgery only" controls.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Courneya, PhD, Principal Investigator — University of Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada